CLINICAL TRIAL: NCT03901950
Title: A Phrase I, Open-label, Multi-center, Non-randomized, Does Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of XNW7201 in Subjects With Advanced Solid Tumors
Brief Title: Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of XNW7201 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNW7201-1-02
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: There will be 5 different doses of the study drug that will be tested. The dose of study drug that you will take will depend on when you enter the research project. The first few participants who enter the research project early will take lower doses of the study drug. Participants entering the research project at a later time will take higher doses of the study drug only if the lower doses that have been tested are well tolerated. You will be closely monitored after you take the study drug.
Masking Description: This is an open-label study. Open-label means that subjects and the study doctor will know exactly what tablets subjects are taking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XNW7201 (Experimental)
  Interventions: Drug: XNW7201 tablets

INTERVENTIONS:
Drug: XNW7201 tablets — A wnt pathway inhibitor

SUMMARY:
The research project is testing this potential new medication for advanced solid tumours. This research project is being done to get more information about the study drug (XNW7201). The study drug is a potential new medication that blocks the activity of a protein found in cancer cells called Wnt. Studies have shown that, in cancer, Wnt is involved in the uncontrolled growth of cancer cells and helping them survive. It is hoped that by blocking the activity of Wnt, the study drug may decrease the growth of cancer cells and their survival. The purpose of this research is to check that the study drug is safe and to see how well it is tolerated in participants with locally advanced or metastatic solid tumours. Another purpose is to find out the highest dose that is well tolerated (called the maximum tolerated dose) and the right dose to use in future clinical research studies with this potential new medication.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who are voluntary to participate in this clinical study, able to understand the study procedure and have signed the informed consent form;

  2. Male or female subjects ≥18 years of age;

  3. Subjects with histologically or cytologically confirmed advanced solid tumors after failure of standard of care, or intolerability to standard of care, or with no standard of care;

  4. ECOG Performance Status of 0 or 1 at both the screening and baseline visits;

  5. Life expectancy ≥12 weeks;

  6. Subjects with at least one measurable lesion in accordance with RECIST 1.1(not required for dose escalation part);

  7. Adequate laboratory parameters during screening as evidenced by:
  * Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L and hemoglobin ≥90 g/dL;
  * Basically normal liver function: total bilirubin ≤ 1.5 × upper limit of normal (ULN); ALT and AST≤2.5 × ULN or ≤ 5 × ULN when metastases to liver occurs;
  * Normal renal function: serum creatinine level>1.5 × ULN or endogenous creatinine clearance <60 mL/min (using Cockcroft-Gault formula);
  * Basically normal coagulation: prothrombin time (PT), international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
  * Cardiac function: left ventricular ejection fraction (LVEF) ≥50%; basically normal ECG, QTcF interval≤70 ms (QTc interval corrected by Fridericia's Correction Formula);

Exclusion Criteria:

* 1. Known or suspected history of allergy to XNW7201 tablet and its metabolite or its excipients;

  2. Subjects who previously received treatment with WNT inhibitor;

  3. Subjects with one of the various factors affecting absorption of oral drugs (e.g., inability to swallow, chronic diarrhoea and intestinal obstruction) or active gastrointestinal disorder, gastric bypass or other diseases that could significantly affect drug absorption, distribution, metabolism or excretion;

  4. Presence of CTCAE Grade > 1 adverse events induced by previous treatment that is still not relieved prior to the first dose, not including alopecia and tolerable adverse event as judged by investigators;

  5. Participation in other clinical studies within 4 weeks prior to the first dose of XNW7201;

  6. Any chemotherapy, biotherapy, radiotherapy, hormone therapy, targeted anti-tumor therapy (excluding nitrosourea and mitomycin C) administered within 4 weeks before the first dose of the investigational drug); nitrosourea or mitomycin C administered within 6 weeks before the first dose of the investigational drug;

  7. Major surgery or active ulcer or incomplete healing of wound within 4 weeks prior to the first dose;

  8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, severe active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent;

  9. Any unstable, pre-existing major medical condition that in the opinion of the investigator contraindicates the use of the investigational drug, including known human immunodeficiency (HIV) or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection;

  10. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of XNW7201 tablets in subjects with advanced solid tumor; | From date of first dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to about 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
The dose-limiting toxicity (DLT) of XNW7201 | At the end of Cycle 1 (each cycle is 30 days)
  Dose-limiting toxicity (DLT) is defined as the adverse events these Grade ≥3 related to XNW7201 treatment that occur from single dose to the last day of Cycle 1 in multiple doses in the dose escalation stage (CTCAE, V5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Le, Study Chair — Evopoint Biosciences Inc.
Locations (1):
- Integrated Clinical Oncology network Pty Ltd, South Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No